CLINICAL TRIAL: NCT01804140
Title: Screening Protocol to Detect BRAF V600 Mutation-Positive Patients for Enrollment Into Clinical Research Studies of Vemurafenib
Brief Title: A Screening Study to Detect BRAF V600 Mutation-Positive Patients For Enrollment Into Clinical Research Studies of Zelboraf (Vemurafenib)
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28560
Record Dates: First submitted 2013-02-26; First posted 2013-03-05 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Myeloma, Neoplasms
MeSH Terms: conditions — Multiple Myeloma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Formalin-fixed paraffin-embedded (FFPE) tumor samples

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This is a screening study to detect BRAF V600 mutation-positive patients for enrollment into clinical research studies of Zelboraf (vemurafenib). Tumor samples will be collected and analyzed from eligible patients with solid tumors (other than metastatic melanoma or papillary thyroid cancer) or multiple myeloma. All institutions with identified patients as defined by this screening protocol will have potential access to the separate vemurafenib protocol MO28072.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumors (excluding melanoma and papillary thyroid cancer) or multiple myeloma refractory to standard therapy or for which standard or curative therapy does not exist or is not considered appropriate by the investigator
* Patients with multiple myeloma must have received at least one line of prior systemic therapy for the treatment of multiple myeloma

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status > 2
* Uncontrolled concurrent malignancy
* Active or untreated CNS metastases
* History of known carcinomatous meningitis
* Prior treatment with a BRAF or MEK inhibitor (prior sorafenib is allowed)
* Uncontrolled, severe medical illness or condition as defined in protocol MO28072

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors (other than metastatic melanoma or papillary thyroid cancer) or multiple myeloma
Sampling Method: Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (18):
- United States (18):
  - Sedona, Arizona
  - Tucson, Arizona
  - Burbank, California
  - Rancho Cucamonga, California
  - Denver, Colorado
  - Ocala, Florida
  - Woodbury, Minnesota
  - Columbia, Missouri
  - Las Vegas, Nevada
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Dallas, Texas
  - Denton, Texas
  - McAllen, Texas
  - Tyler, Texas
  - Spokane, Washington
  - Yakima, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Confirmed Solid Tumors or Multiple Myeloma: Participants with solid tumors (other than metastatic melanoma or papillary thyroid cancer) or multiple myeloma who met the inclusion criteria and did not meet exclusion criteria of the study were enrolled and were evaluated for the presence of BRAF V600 mutations by collecting tumor samples or performing fresh biopsies according to local standards.
Period: Overall Study
Arm/Group | Participants With Confirmed Solid Tumors or Multiple Myeloma
Started | 662 (This includes all the participants who were enrolled for this study.)
Completed | 548 (This includes all the participants with mutation results from the sampling or biopsy procedures.)
Not Completed | 114
Not completed — No sampling or biopsy procedures done | 114

BASELINE CHARACTERISTICS:
Population: All the participants who were enrolled and were evaluable for the BRAF V600 mutations were included in the analysis.
Arm/Group | Participants With Confirmed Solid Tumors or Multiple Myeloma
Number analyzed (Participants) | 548
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (12.38)
Gender [Count of Participants; unit: Participants]
  Female | 326
  Male | 222

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With BRAF V600 Mutation Positivity in Tumor Samples by Cancer Type
Description: Formalin-fixed paraffin-embedded (FFPEs) tumor samples (at least 5 serially-cut, unstained, 5 micrometer [μm] sections) were collected from eligible participants who consented to participate in the study. FFPE tumor samples were either from archived sections (from the initial diagnosis of cancer) or from fresh biopsies that were performed according to local standards. Tumor samples were then sent to a central laboratory to identify activating BRAF V600 mutations. Identification of mutations was done using bidirectional direct Sanger sequencing procedure.
Time Frame: Up to 1 year
Population: All the participants who were enrolled and were evaluable for the BRAF V600 mutations were included in the analysis. n is the number of participants with that type of cancer in the total population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With Confirmed Solid Tumors or Multiple Myeloma
Number analyzed (Participants) | 548
percentage of participants
  Breast cancer (n=85) | 0 [0 to 0]
  Non-small cell lung carcinoma (n=65) | 3 [0.4 to 10.7]
  Colorectal cancer (n=74) | 11 [4.8 to 20.2]
  Ovarian cancer (n=66) | 0 [0 to 0]
  Prostate cancer (n=21) | 0 [0 to 0]
  Multiple myeloma (n=31) | 3 [0.1 to 16.7]
  Biliary tract cancer (n=16) | 6 [0.2 to 30.2]
  Other cancer (n=190) | 2 [0.6 to 5.3]
  Overall (n=540) | 3 [1.7 to 4.7]

2. Primary Outcome: Number of Participants Classified Based on Different Types of BRAF V600 Mutation Patterns in Tumor Samples
Description: FFPEs tumor samples (at least 5 serially-cut, unstained, 5 μm sections) were collected from eligible participants who consented to participate in the study. FFPE tumor samples were either from archived sections (from the initial diagnosis of cancer) or from fresh biopsies that were performed according to local standards. Tumor samples were then sent to a central laboratory to identify activating BRAF V600 mutations. Identification of mutations was done using bidirectional direct Sanger sequencing procedure. V600E, V600K, V600D, and V600R are the different types of BRAF V600 mutations.
Time Frame: Up to 1 year
Population: All the participants who were enrolled and were evaluable for the BRAF V600 mutations were included in the analysis.
Measure: Number; unit: participants
Arm/Group | Participants With Confirmed Solid Tumors or Multiple Myeloma
Number analyzed (Participants) | 548
participants
  BRAF V600E | 16
  BRAF V600K | 0
  BRAF V600D | 0
  BRAF V600R | 0
  Other V600 | 0

ADVERSE EVENTS:
Time Frame: All adverse events that occurred up to 28 days after the biopsy was performed or those adverse events that the physician considered to have causal relationship to the biopsy performed were recorded.
Arm/Group | Participants With Confirmed Solid Tumors or Multiple Myeloma
Serious Adverse Events (participants affected / at risk) | 0/548
Other Adverse Events (participants affected / at risk) | 0/548

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.